CLINICAL TRIAL: NCT02460068
Title: A Randomized, Phase III Study of Fotemustine Versus the Combination of Fotemustine and Ipilimumab or the Combination of Ipilimumab and Nivolumab in Patients With Metastatic Melanoma With Brain Metastasis
Brief Title: A Study of Fotemustine(FTM) Vs FTM and Ipilimumab (IPI) or IPI and Nivolumab in Melanoma Brain Metastasis
Acronym: NIBIT-M2
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Italian Network for Tumor Biotherapy Foundation (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NIBIT-M2
Record Dates: First submitted 2015-05-22; First posted 2015-06-02 (Estimated); Last update posted 2015-06-02 (Estimated); Status verified 2015-05

CONDITIONS: Brain Metastases
Keywords: melanoma brain metastases; nivolumab; ipilimumab
MeSH Terms: conditions — Brain Neoplasms | interventions — fotemustine; Ipilimumab; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- fotemustine (Active Comparator): fotemustine alone
  Interventions: Drug: Fotemustine
- fotemustine and ipilimumab (Experimental): fotemustine in combination with ipilimumab
  Interventions: Drug: Fotemustine and Ipilimumab
- ipilimumab and nivolumab (Experimental): ipilimumab in combination with nivolumab
  Interventions: Drug: Ipilimumab and nivolumab

INTERVENTIONS:
Drug: Fotemustine — Fotemustine: fotemustine at 100 mg/mq intravenously (i.v.) over 60 minutes once every week for 3 doses, and once every 3 weeks from week 9 for 6 doses.
  Other Names: Fotemustine (Muphoran);
  Arms: fotemustine
Drug: Fotemustine and Ipilimumab — Fotemustine and ipilimumab:fotemustine 100 mg/m2 i.v. over 60 minutes once every week for 3 weeks (Weeks 1, 2, 3) plus ipilimumab at 10 mg/kg i.v. over 90 minutes every 3 weeks for 4 cycles (Weeks 1, 4, 7, 10); fotemustine 100 mg/m2 i.v. over 60 minutes once every 3 weeks from week 9 for 6 doses plus ipilimumab at 10 mg/kg i.v. over 90 minutes every 12 weeks from week 24.
  Other Names: Fotemustine (Muphoran);; Ipilimumab (YERVOY)
  Arms: fotemustine and ipilimumab
Drug: Ipilimumab and nivolumab — ipilimumab and nivolumab: ipilimumab 3 mg/kg i.v over 90 minutes combined with nivolumab 1 mg/kg i.v over 60 minutes every three weeks for 4 doses, then nivolumab 3 mg/kg IV over 60 minutes every two weeks.
  Other Names: Ipilimumab (YERVOY); Nivolumab (OPDIVO)
  Arms: ipilimumab and nivolumab

SUMMARY:
This Phase 3, open-label, triple arm study aims to evaluate the overall survival (OS) of fotemustine versus the combination of ipilimumab and fotemustine or the combination of Ipilimumab and nivolumab in patients with metastatic melanoma with brain metastasis.

DETAILED DESCRIPTION:
Metastatic melanoma is an aggressive tumor associated with very poor prognosis. Brain metastases develop in nearly half of MM pts and in 30 to 40% of these subjects, the brain is the first site of relapse. The limited activity of available agents, along with relative resistance to radiotherapy and poor CNS penetration of most chemotherapeutic agents, make this one of the most daunting problems in oncology. There is no optimal systemic or local therapy for melanoma metastatic to the brain. Though MM pts with brain metastases have been excluded from most phase II-III trials with ipilimumab, initial evidences suggest that the anti-CTLA-4 monoclonal antibody ipilimumab might be active as single-agent also in this clinical setting. Preliminary results from the NIBIT-M1 phase II trial suggest for the safety and efficacy of the combination of fotemustine plus ipilimumab in MM pts with or w/o brain metastases.Recent data from a phase I study in MM pts w/o brain metastases have shown that concurrent administration of ipilimumab (3 mg/kg) plus the anti-PD1 mAb nivolumab (1 mg/kg) induced objective responses in 53% of pts, with a tumor reduction of ≥80% in 41% of pts, with an 82% 1-year OS, and with an acceptable safety profile.Based on the long-term follow-up of the NIBIT-M1 study, and on the activity of the concurrent administration of ipilimumab and nivolumabthe NIBIT-M2 study will explore the efficacy of the combination of ipilimumab and fotemustine or ipilimumab and nivolumab versus fotemustine alone in pts with melanoma metastatic to the brain.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to give written informed consent.
* Histologic diagnosis of malignant melanoma;
* Stage IV melanoma;
* No prior therapy for advanced (unresectable Stage III or Stage IV) disease;
* No previous systemic corticosteroid therapy within 7 days;
* Prior adjuvant treatment with IFN or other immunotherapy allowed with exception of anti-CTLA-4;
* Presence of asymptomatic brain metastases: patients must have measurable metastases in the brain, defined as lesions that can be accurately measured in 2 dimensions as ≥ 0.5 cm (maximum 2 cm) in the brain MRI with contrast;
* Pts who have been previously treated with brain stereotactic radiotherapy (SRT), whole-brain radiotherapy (WBRT) and/or surgery, must have developed new measurable brain lesions;
* Life expectancy ≥ 12 weeks;
* ECOG performance status of 0 or 1 (see Appendix 2);
* Normal laboratory tests were required.
* Subjects must have known BRAF V600E mutation status or consent to BRAF V600E mutation testing per local institutional standard.
* Negative screening tests for HIV, Hepatitis B, and Hepatitis C.
* Men and women, of and over 18 years old.Women of childbearing potential (WOCBP) must use appropriate method(s) of contraception. WOCBP should use an adequate method to avoid pregnancy for 23 weeks (30 days plus the time required for nivolumab to undergo five half-lives) after the last dose of investigational drug

Exclusion Criteria:

* Any malignancy from which the patient has been disease-free for less than 5 years, with the exception of adequately treated and cured basal or squamous cell skin cancer, superficial bladder cancer, carcinoma in situ of the cervix;
* Primary ocular or mucosal melanoma.

Medical History and Concurrent Diseases:

* Symptomatic brain metastases requiring immediate local intervention (radiotherapy (RT) and/or surgery);
* Autoimmune disease
* Any underlying medical condition, which in the opinion of the investigator, will make the administration of study drug hazardous or obscure the interpretation of adverse events, such as a condition associated with frequent diarrhea.

Prohibited Treatments and/or Therapies:

* Concomitant therapy with any anti-cancer agent; immunosuppressive agents; any non-oncology vaccine therapy used for prevention of infectious diseases (for up to 1 month prior to or after any dose of study drug); surgery or radiotherapy ; other investigational anti-cancer therapies; or chronic use of systemic corticosteroids
* Previous treatment with other investigational products, including cancer immunotherapy, within 30 days;
* Prior treatment with anti-CTLA-4 and/or , anti-PD1/PD-L1 or fotemustine.

Sex and Reproductive Status:

* WOCBP who are unwilling or unable to use an acceptable method to avoid pregnancy for the entire study period and for up to 8 weeks after the study;
* Women who are pregnant or breastfeeding;
* Women with a positive pregnancy test on enrollment or prior to investigational product administration;
* Sexually active fertile men not using effective birth control if their partners are WOCBP.

Other Exclusion Criteria:

* Prisoners or subjects who are involuntarily incarcerated;
* Subjects who are compulsorily detained for treatment of either a psychiatric or physical illness.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 168 (Estimated)
Dates: Start 2012-12; Primary Completion 2018-01 (Estimated); Study Completion 2020-01 (Estimated)

PRIMARY OUTCOMES:
Overall Survival (OS) | 2 years
  To compare the efficacy of the combination of ipilimumab and fotemustine or the Combination of ipilimumab and nivolumab versus fotemustine in terms of overall survival (OS) in patients with metastatic melanoma with brain metastasis.Overall Survival (OS) is defined as the time from randomization until the date of death. For those subjects who have not died, OS will be censored at the recorded last date of subject contact, and for subjects with a missing recorded last date of contact, OS will be censored at the last date the subject was known to be alive.

SECONDARY OUTCOMES:
safety (adverse events) | 2 years
  Reporting of safety, extent of exposure, concomitant medications and discontinuation of study therapy will be based on all treated subjects; for on-study laboratory test results, all treated subjects with at least one on-study laboratory measurement available will be included in the analysis. The reporting period for safety data will be from the date of first dose received on this study to 70 days (5 half-lives) after the last dose is received. Serious adverse events are reported from the time of consent forward for all subjects.All subjects who receive at least 1 dose of study treatment will be evaluated for safety parameters
m-WHO and immune-related Disease Control Rate (DCR) in and outside the brain | Weeks 24
  m-WHO and immune-related is the proportion of treated subjects with a ir-BOR of confirmed irCR, confirmed irPR or irSD in and outside the brain.
Immune-related Progression-free Survival (irPFS) | 2 years
  Immune-related progression free survival (irPFS) per irRC will be defined as the time between the date of randomization and the date of progression per irRC or death, whichever occurs first. A subject who dies without reported progression per irRC will be considered to have progressed on the date of death.
m-WHO Progression-free Survival (irPFS) | 2 years
  Progression-free survival (PFS) per mWHO criteria will be defined as the time between the date of randomization and the date of progression per mWHO criteria or death, whichever occurs first. A subject who dies without reported progression per mWHO criteria will be considered to have progressed on the date of death.
Objective Response Rate (ORR) | Weeks 24
  is the proportion of treated subjects with a BOR of confirmed CR or confirmed PR.
Immune-related Objective Response Rate (irORR) | Weeks 24
  is the proportion of treated subjects with a irBOR of confirmed irCR or confirmed irPR.
Time to Response (TTR) | Weeks 24
  Time to Response (TTR) is defined as the time from first dosing date until the measurement criteria are first met for overall response of PR or CR (whichever status comes first, and provided it is subsequently confirmed).
Immune-related Time to Response (irTTR) | Weeks 24
  Immune-related Time to Response (irTTR) is defined as the time from first dosing date until the measurement criteria are first met for overall response of irPR or irCR (whichever status comes first, and provided it is subsequently confirmed).
Duration of Response (DoR) | 2 years
  Duration of Response (DoR) is defined as the time between the date the measurement criteria are first met for an CR or PR (whichever status comes first and provided it is subsequently confirmed) and the date of PD or death (whichever comes first). For a subject who undergoes tumor resection following response but prior to disease progression, DOR will be censored at the date of the last evaluable TA on or prior to the date of resection. For subjects who remain alive and have no progressive disease as assessed by the investigator using RC, DOR will be censored on the date of last evaluable tumor assessment.
Immune-related Duration of Response (irDoR) | 2 years
  Immune-related Duration of Response (irDoR) for the subjects whose irBOR is irCR or irPR will be defined as the time between the date of response of confirmed irCR or confirmed irPR (whichever occurs first) and the date of irPD or death (whichever occurs first). The onset of a confirmed irCR or irPR is determined by the initial assessment of response, not by the confirmatory assessment. Note that if an assessment of irPR occurs before confirmation of irCR, the duration of immune-related response endpoint will not begin at the time that the irBOR of irCR is shown but rather at the earlier time-point showing irPR. For subjects who remain alive and have not progressed following response, irDoR will be censored on the date of last evaluable TA.
Brain progression-free survival (Brain-PFS) | 6 months
  Brain progression-free survival (Brain-PFS) (3 and 6 months rates) is defined as the time from randomization date to the date of progression as per MRI of existing brain lesions, or of occurrence as per MRI of a new lesion located in the brain, or of death, whichever occurs first. For subjects who remain alive and have not progressed as per definition above, Brain-PFS will be censored at the day of last evaluable brain imaging assessment.

CONTACTS AND LOCATIONS:
Overall Officials: Anna Maria Di Giacomo, PhD,MD, Principal Investigator — Medical Oncology and Immunotherapy Unit, University Hospital of Siena
Locations (11):
- Italy (11):
  - Medical Oncology, Cancer Institute "Giovanni Paolo II", Bari
  - Medical Oncology, Pope Giovanni XXIII Hospital, Bergamo
  - National Institute for Cancer Research, Genoa
  - Immunotherapy and Somatic Cell Therapy Unit, Scientific Institute of Romagna, Meldola
  - Surgical Oncology, National Cancer Institute, Milan
  - European Institute of Oncology, Milan
  - Medical Oncology and Innovative Therapy, National Cancer Institute, Naples
  - esophageal and melanoma oncology, Istituto Oncologico Veneto, Padua
  - Medical Oncology, National Cancer Institute "Regina Elena", Rome
  - Medical Oncology and Immunotherapy Unit, University Hospital of Siena, Siena
  - S C Dermatology, A.O.U. City of Health and Science of Turin, Turin

REFERENCES:
- [Background] Avril MF, Aamdal S, Grob JJ, Hauschild A, Mohr P, Bonerandi JJ, Weichenthal M, Neuber K, Bieber T, Gilde K, Guillem Porta V, Fra J, Bonneterre J, Saiag P, Kamanabrou D, Pehamberger H, Sufliarsky J, Gonzalez Larriba JL, Scherrer A, Menu Y. Fotemustine compared with dacarbazine in patients with disseminated malignant melanoma: a phase III study. J Clin Oncol. 2004 Mar 15;22(6):1118-25. doi: 10.1200/JCO.2004.04.165. PMID 15020614
- [Background] Margolin K, Ernstoff MS, Hamid O, Lawrence D, McDermott D, Puzanov I, Wolchok JD, Clark JI, Sznol M, Logan TF, Richards J, Michener T, Balogh A, Heller KN, Hodi FS. Ipilimumab in patients with melanoma and brain metastases: an open-label, phase 2 trial. Lancet Oncol. 2012 May;13(5):459-65. doi: 10.1016/S1470-2045(12)70090-6. Epub 2012 Mar 27. PMID 22456429
- [Background] Di Giacomo AM, Ascierto PA, Pilla L, Santinami M, Ferrucci PF, Giannarelli D, Marasco A, Rivoltini L, Simeone E, Nicoletti SV, Fonsatti E, Annesi D, Queirolo P, Testori A, Ridolfi R, Parmiani G, Maio M. Ipilimumab and fotemustine in patients with advanced melanoma (NIBIT-M1): an open-label, single-arm phase 2 trial. Lancet Oncol. 2012 Sep;13(9):879-86. doi: 10.1016/S1470-2045(12)70324-8. Epub 2012 Aug 13. PMID 22894884
- [Background] Di Giacomo AM, Ascierto PA, Queirolo P, Pilla L, Ridolfi R, Santinami M, Testori A, Simeone E, Guidoboni M, Maurichi A, Orgiano L, Spadola G, Del Vecchio M, Danielli R, Calabro L, Annesi D, Giannarelli D, Maccalli C, Fonsatti E, Parmiani G, Maio M. Three-year follow-up of advanced melanoma patients who received ipilimumab plus fotemustine in the Italian Network for Tumor Biotherapy (NIBIT)-M1 phase II study. Ann Oncol. 2015 Apr;26(4):798-803. doi: 10.1093/annonc/mdu577. Epub 2014 Dec 23. PMID 25538176
- [Background] Wolchok JD, Kluger H, Callahan MK, Postow MA, Rizvi NA, Lesokhin AM, Segal NH, Ariyan CE, Gordon RA, Reed K, Burke MM, Caldwell A, Kronenberg SA, Agunwamba BU, Zhang X, Lowy I, Inzunza HD, Feely W, Horak CE, Hong Q, Korman AJ, Wigginton JM, Gupta A, Sznol M. Nivolumab plus ipilimumab in advanced melanoma. N Engl J Med. 2013 Jul 11;369(2):122-33. doi: 10.1056/NEJMoa1302369. Epub 2013 Jun 2. PMID 23724867
- See also: Fondazione NIBIT — http://www.fondazionenibit.org/